CLINICAL TRIAL: NCT04110873
Title: A Phase II, Three-arms, Double-blind, Dosing-ranging, Placebo-controlled Trial Evaluating the Efficacy of Antroquinonol in Patients With Atopic Dermatitis
Brief Title: A Phase II, Placebo-controlled Trial Evaluating the Efficacy of Antroquinonol in Patients With Atopic Dermatitis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: It was hard to find suitable subject due to strict enrollment criteria.
Sponsor: Chung Shan Medical University (Other)
Collaborators: Golden Biotechnology Corporation (Industry)
Responsible Party: Principal Investigator, Cheng-Chung Wei, Chung Shan Medical University Hospital, Chung Shan Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CS17155
Record Dates: First submitted 2019-09-30; First posted 2019-10-01 (Actual); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Atopic Dermatitis
Keywords: antroquinonol, Atopic dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — antroquinonol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Antroquinonol capsule 50mg (Experimental): patients will receive Antroquinonol 50mg per day (QD) on Day 1 for 12 weeks
  Interventions: Drug: Antroquinonol Capsule 50mg
- Antroquinonol capsule 100mg (Experimental): patients will receive Antroquinonol 100mg per day (QD) on Day 1 for 12 weeks
  Interventions: Drug: Antroquinonol Capsule 100mg
- Placebo oral capsule (Placebo Comparator): patients will receive placebo per day (QD) on Day 1 for 12 weeks
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: Antroquinonol Capsule 50mg — patients will receive Antroquinonol 50mg per day (QD) on Day 1 for 12 weeks
  Other Names: Antroquinonol 50mg
  Arms: Antroquinonol capsule 50mg
Drug: Antroquinonol Capsule 100mg — patients will receive Antroquinonol 100mg per day (QD) on Day 1 for 12 weeks
  Other Names: Antroquinonol 100mg
  Arms: Antroquinonol capsule 100mg
Drug: Placebo oral capsule — patients will receive placebo per day (QD) on Day 1 for 12 weeks
  Other Names: Placebo
  Arms: Placebo oral capsule

SUMMARY:
Primary Objective:

To evaluate the activity of Antroquinonol in patients with atopic dermatitis.

Secondary Objective:

To assess the mechanism and cytokines change of Antroquinonol in patients with atopic dermatitis.

Exploratory Objective:

To explore potential relationships between Antroquinonol exposure and safety and efficacy endpoints.

DETAILED DESCRIPTION:
This is a Phase II, three-arms, double-blind, dosing-ranging, placebo-controlled trial evaluating the efficacy of Antroquinonol in patients with atopic dermatitis. The study is conducted in compliance with the guidelines for Good Clinical Practice and the Declaration of Helsinki. Approval is obtained from the local ethics committee or institutional review board at each study center. All the patients provided written informed consent.

60 patients totally (20 patients per arm) with atopic dermatitis will receive Antroquinonol or placebo. A patient will have received at one dose of Antroquinonol or placebo with tropical urea ointment and have three baseline scores assessment (see Statistical Methods). Enrollment will continue until the target number of evaluable patients has been enrolled.

Written informed consent must be obtained from all patients before initiating Screening. The Screening period will be up to 14 days in duration (Days -14 to -1). Following completion of all Screening assessments and confirmation of eligibility criteria, patients will receive Antroquinonol 50mg, 100mg or placebo per day (QD) on Day 0 for 12 weeks or until documented evidence of unacceptable toxicity, non-compliance or withdrawal of consent by the patient, or the investigator decides to discontinue treatment, whichever comes first. The time of study drug administration should be recorded in the patient diary.

Patients will attend study visits on Days 0, 28, 56 and 84. The following procedures will be performed according to the schedule of assessments: physical examination, vital signs, performance status, clinical laboratory tests, adverse events (AEs), concomitant medication and patient compliance.

Scores assessments will be performed at Screening, Day 28, Day 56 and Day 84 including EASI score, SCORAD, sIGA score, BSA affected by atopic dermatitis and pruritus verbal rating scale.

The primary endpoint is the percentage improvement between baseline and week 12 in Eczema Area and Severity Index (EASI).

ELIGIBILITY:
Inclusion Criteria:

1. Patients between the ages of 20 and 65 years who had moderate-to-severe atopic dermatitis (using the Hanifin and Rajka Diagnostic Criteria)
2. Patients with body weight ≥ 25 kg and ≤ 120 kg, signing informed consent
3. To be eligible to participate, patients were required to have

   1. a score of at least 5 on the Eczema Area and Severity Index (EASI), which ranges from 0 to 72, with higher scores indicating worse disease severity;
   2. a score for pruritus of at least 30 mm on a visual-analogue scale, which ranges from 0 (no itch) to 100 mm (worst itch imaginable);
   3. a score of at least 2 on the static Investigator's Global Assessment (sIGA), which ranges from 0 (clear) to 4 ( severe disease).
   4. BSA affected or PSAI ≥ 5%

Exclusion Criteria:

Patients meeting any of the following criteria must not be enrolled in the study:

1. Patients with active dermatologic diseases concomitant with atopic dermatitis.
2. Patients with severe medical condition(s) that in the view of the investigator prohibits participation in the study
3. Subjects with defective epidermal barrier(e.g Netherton's syndrome)
4. Any subject who is immunocompromised or has a history of malignant disease. This information will be gathered verbally from the patient while taking a medical history from the patient, and will not involve further testing such as an HIV test.
5. Subjects with a history of psychiatric disease or history of alcohol or drug abuse that would interfere with the ability to comply with the study protocol
6. Any noticeable breaks or cracks in the skin on either arm, including severely excoriated skin or skin with open or weeping wounds suggestive of an active infection or increased susceptibility to infection.
7. Ongoing participation in another investigational trial
8. Use of any oral or topical antibiotic for up to four weeks prior to the Treatment visit or active infection that in the opinion of the investigator would compromise the patient's ability to tolerate therapy
9. Use of any systemic immunosuppressive therapy (e.g. CsA, MTX, etc.) within four weeks of the Treatment visit.
10. Participant who has a condition or is in a situation that, in the investigator's opinion, may put the patient at significant risk, or may significantly interfere with the patient's participation in the study.
11. Subjects with prosthetic heart valves, pacemakers, intravascular catheters, or other foreign or prosthetic devices.
12. History of food or drug-related severe anaphylactoid or anaphylactic reaction(s)
13. Pregnancy or breastfeeding
14. History or presence of epilepsy, significant neurological disorders, cerebrovascular attack or ischemia
15. History or presence of myocardial infarction or cardiac arrhythmia under drug therapy
16. Patients who are unable to complete questionnaires on paper.
17. Clinically significant laboratory abnormalities.
18. History of malignancy of any organ system, treated or untreated.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2018-07-27 (Actual); Primary Completion 2019-06-25 (Actual); Study Completion 2019-06-25 (Actual)

PRIMARY OUTCOMES:
Eczema Area and Severity Index (EASI) | week 0(baseline) and week12
  The percentage improvement between week 0(baseline) and week 12 in Eczema Area and Severity Index (EASI)

SECONDARY OUTCOMES:
Eczema Area and Severity Index (EASI) at each time point | week 0(baseline), week 4, week8 and week12
  Secondary endpoints at week 12 and at each time point (weeks 4, 8 and 12) included improvement from baseline in the EASI score
Scoring Atopic Dermatitis (SCORAD) | week 0(baseline), week 4, week8 and week12
  Secondary endpoints at week 12 and at each time point (weeks 4, 8 and 12) included improvement from baseline in the Scoring Atopic Dermatitis (SCORAD), which ranges from 0 to 103, with higher scores indicating more severe disease
static Investigator's Global Assessment (sIGA) | week 0(baseline), week 4, week8 and week12
  Secondary endpoints at week 12 and at each time point (weeks 4, 8 and 12) included improvement from baseline in the sIGA score
Body-surface area affected by atopic dermatitis | week 0(baseline), week 4, week8 and week12
  Secondary endpoints at week 12 and at each time point (weeks 4, 8 and 12) included improvement from baseline in the Body-surface area affected by atopic dermatitis
Pruritus verbal rating scale | week 0(baseline), week 4, week8 and week12
  Secondary endpoints at week 12 and at each time point (weeks 4, 8 and 12) included improvement from baseline in the Pruritus verbal rating scale, which describes pruritus intensity from 0 (none) to 10(very severe) daily
Sleep-disturbance visual-analogue scale | week 0(baseline), week 4, week8 and week12
  Secondary endpoints at week 12 and at each time point (weeks 4, 8 and 12) included improvement from baseline in the Sleep-disturbance visual-analogue scale, which ranges from 0 (no sleep disturbance) to 10 (inability to sleep at all) daily
The proportion of patients with 25%, 50%, and 75% improvement in scores on the pruritus visual-analogue scale | week 0(baseline), week 4, week8 and week12
  Secondary endpoints at week 12 and at each time point (weeks 4, 8 and 12) included improvement from baseline in the proportion of patients with 25%, 50%, and 75% improvement in scores on the pruritus visual-analogue scale
The proportion of patients with 25%, 50%, and 75% improvement in scores on the EASI | week 0(baseline), week 4, week8 and week12
  Secondary endpoints at week 12 and at each time point (weeks 4, 8 and 12) included improvement from baseline in the proportion of patients with 25%, 50%, and 75% improvement in scores on the EASI
The proportion of patients with 25%, 50%, and 75% improvement in scores on the SCORAD | week 0(baseline), week 4, week8 and week12
  Secondary endpoints at week 12 and at each time point (weeks 4, 8 and 12) included improvement from baseline in the proportion of patients with 25%, 50%, and 75% improvement in scores on the SCORAD
The proportion of patients with an improvement of at least 2 points on the sIGA | week 0(baseline), week 4, week8 and week12
  Secondary endpoints at week 12 and at each time point (weeks 4, 8 and 12) included improvement from baseline in the proportion of patients with an improvement of at least 2 points on the sIGA
The proportion of patients with an improvement of at least 2 points on the pruritus verbal rating scale | week 0(baseline), week 4, week8 and week12
  Secondary endpoints at week 12 and at each time point (weeks 4, 8 and 12) included improvement from baseline in the proportion of patients with an improvement of at least 2 points on the pruritus verbal rating scale

OTHER OUTCOMES:
The percentage change between baseline and week 12 in serum cytokines | week 0(baseline) and week12
  The percentage change between baseline and week 12 in serum cytokines:
  TARC/CCL17, IFN-gamma, TNF-alpha, IL-18, IL-6, IL-1beta

CONTACTS AND LOCATIONS:
Overall Officials: Wei C- C, M.D., Principal Investigator — Chung Shan Medical University
Locations (1):
- Chung Shan Medical University Hospital, Taichung, Taiwan